CLINICAL TRIAL: NCT02400684
Title: ENDmetriosis and Reserve Ovarienne
Acronym: ENDRO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6017
Record Dates: First submitted 2015-03-23; First posted 2015-03-27 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2015-09

CONDITIONS: Deep Endometriosis Stage III; Deep Endometriosis Stage IV
Keywords: AFSr classification; laparoscopy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 3 times blood sample retrieval and use serum to measure AMH the primary end point but also FSH, LH, estradiol which are study usually.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Deep endometriosis: The population is a female population, above 18 years and under 38 years who have stage III or IV endometriosis (which will remain to be confirmed after inclusion by intra-operative observations), and who undergo operative laparoscopy in our center, with only deep endometriosis without endometriomas.
  Interventions: Biological: blood samples
- Deep endometriosis and endométriomas: The population is a female population, above 18 years and under 38 years who have stage III or IV endometriosis (which will remain to be confirmed after inclusion by intra-operative observations), and who undergo operative laparoscopy in our center, with deep endometriosis and endometriomas.
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — Evolution of AMH before and after deep endometriosis surgery

SUMMARY:
Endometriosis is the ectopic implantation of endometrial glands and stroma, and can be ovarian and peritoneal (superficial or deep). There are 4 stages in endometriosis according to severity, and the stage is established on the basis of intra-operative observations. The AFSr classification is currently most used (I-IV,minimal, mild, moderate, severe). Most associated with endometriosis are subfertility and pelvic pain.

In the surgical management of deep endometriosis, the issue of fertility is pivotal. There is a higher rate of infertility in a population of women with endometriosis as compared to the general population, even though the mechanisms are not yet elucidated. Patients with deep endometriosis can be referred to the surgeon for subfertility, but even when they are referred for chronic pain, future fertility considerations are taken into account in the planning of the surgery, as the patients are often young.

It is now well documented that ovarian cystectomy is deleterious with regards to the ovarian reserve, and more so in endometriomas than in any other type of benign cysts. The ovarian reserve is the functional potential of the ovaries, reflecting the quantity and quality of remaining follicles. Studies have also relied greatly on the measure of serum anti-mullerian hormone (AMH) to evaluate the effect of cystectomy on ovarian reserve, as AMH is currently the most reliable marker to assess ovarian reserve. A significant difference was found between AMH before and following cystectomy in several studies. The deleterious effect of deep endometriosis surgery which comprises a wide dissection and adhesiolysis of the pelvis in many cases, even when no cystectomy has been performed, is therefore not entirely ruled out. To the best of our knowledge, there are no studies on the effect of deep endometriosis surgery, apart from ovarian surgery, on ovarian reserve.

Our center is very active in the laparoscopic surgical treatment of deep endometriosis, with more than 200 cases every year. The objective of this trial is to assess the effect of deep endometriosis surgery on the ovarian reserve, whether a cystectomy is performed or not, by measuring serum AMH before and after surgery, at 6 months and 1 year post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* female patient between 18 and 38 years
* endometriosis stage III or IV in the AFSr classification
* laparoscopy included deep endometriosis procedures (adhesiolysis, ureterolysis, cystectomy, resection of bowel, urinary or deep peritoneal endometriosis)
* written informed consent

Exclusion Criteria:

* previous adnexectomy or adnexectomy during surgery

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female between 18 and 38 years old Deep endometriosis stage III or IV endometriosis of AFSr classification who undergo laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2015-06; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ovarian reserve (determined by AMH) at one year | Baseline : before surgery (less than one month) and one year after surgery

SECONDARY OUTCOMES:
Percentage of decline in AMH between patients who underwent ovarian cystectomy and those who did not | baseline and 1 year after surgery
Evolution curve of AMH at 6 months and 1 year post-operatively | baseline, 6 months and 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine RONGIERES, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - CMCO - Hôpitaux Universitaires de Strasbourg, Schiltigheim
  - Hôpital de Hautepierre - Hôpitaux Universitaires de Strasbourg, Strasbourg